CLINICAL TRIAL: NCT03798366
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Efficacy, Safety, and Tolerability of Orally Administered GLPG1690 for 24 Weeks in Subjects With Systemic Sclerosis
Brief Title: A Clinical Study to Test How Effective and Safe GLPG1690 is for Participants With Systemic Sclerosis
Acronym: NOVESA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG1690-CL-204; 2018-001817-33 (EudraCT Number)
Record Dates: First submitted 2019-01-03; First posted 2019-01-09 (Actual); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — GLPG1690

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GLPG1690 600 mg (Experimental): Participants received GLPG1690 600 milligrams (mg), orally once daily for 24 weeks.
  Interventions: Drug: GLPG1690
- Placebo (Placebo Comparator): Participants received GLPG1690 matching placebo, orally once daily for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLPG1690 — Film-coated tablets of GLPG1690 for oral use.
  Arms: GLPG1690 600 mg
Drug: Placebo — Film-coated tablets of GLPG1690 matching placebo for oral use.
  Arms: Placebo

SUMMARY:
The main purpose of the study is to see if GLPG1690 helps (together with the standard of care treatment) in the treatment of the skin and other areas affected by systemic sclerosis.

Another aim is to find out how safe/well tolerated GLPG1690 will be and whether there are any side effects. The study will also look at other things, including whether the study drug affects disease progression and also if it changes any aspect of the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with the protocol requirements and to sign the informed consent form (ICF) as approved by the Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to any screening evaluations.
* Male and female participants ≥18 years at the time of consent who meet the American College of Rheumatology (ACR)/EULAR 2013 diagnostic criteria for systemic sclerosis with diffuse cutaneous involvement (according to LeRoy's criteria) and ≤5 years since the onset of the first systemic sclerosis manifestation other than Raynaud's phenomenon.
* Modified Rodnan Skin Score (mRSS) >10 at screening.
* Active disease at screening, as defined by: Worsening of skin thickening (≥2 mRSS points) as assessed by mRSS measured at screening versus a previous mRSS assessment made within 6 months prior to screening, or new areas of skin involvement within 6 months prior to screening as documented by physician note, or new-onset systemic sclerosis with symptoms or signs other than Raynaud's phenomenon within 2 years prior to screening, or ≥1 tendon friction rub (palpated in the finger flexors or extensors, wrist flexors or extensors, olecranon bursa, shoulders, knees, anterior or posterior ankles with active motion).
* Participant must be able and willing to comply with restrictions on prior and concomitant medication as described in the protocol
* Female participants of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at the baseline visit.
* Female participants of childbearing potential or male participants with female partners of childbearing potential must be willing to comply with the contraceptive methods described in the protocol prior to the first dose of the investigational medicinal product (IMP), during the clinical study, and for at least 90 days after the last dose of the IMP for male participants and 30 days after the last dose of the IMP for female participants.
* A body mass index (BMI) between 18-35 kg/m^2, inclusive, at screening.
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and fasting clinical laboratory safety tests. Clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered non-clinically significant in the opinion of the investigator.

Exclusion Criteria:

* Known hypersensitivity to IMP ingredients or history of a significant allergic reaction to any drug as determined by the investigator, such as anaphylaxis requiring hospitalization.
* Breastfeeding female or participant intending to become pregnant or breastfeed.
* History of or a current immunosuppressive condition (e.g. human immunodeficiency virus [HIV] infection, congenital, acquired).
* Positive blood testing for hepatitis B surface antigen or hepatitis C virus (antibody, confirmed by hepatitis C virus ribonucleic acid [RNA] positivity). Note: Participants with a resolved hepatitis A at least 3 months prior to screening can be screened.
* History of malignancy within the past 5 years (except for carcinoma in situ of the uterine cervix, basal cell carcinoma of the skin that has been treated with no evidence of recurrence, prostate cancer medically managed through active surveillance or watchful waiting, and squamous cell carcinoma of the skin if fully resected and ductal carcinoma in situ).
* Clinically significant abnormalities, in the opinion of the investigator, detected on ECG at screening of either rhythm or conduction, QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 ms, or a known long QT syndrome.
* Unstable cardiovascular, pulmonary, or other disease (other than systemic sclerosis-related), in the opinion of the investigator, within 6 months prior to the baseline visit (e.g. coronary heart disease, heart failure, stroke).
* Severe pulmonary disease with forced vital capacity (FVC) ≤45% of predicted within 6 months prior to the baseline visit.
* Chronic or ongoing active infectious disease, including tuberculosis (requiring hospitalization or systemic treatment within 4 weeks prior to the baseline visit).
* Abnormal liver function test (LFT) at screening, defined as aspartate aminotransferase (AST), and/or alanine aminotransferase (ALT), and/or bilirubin, and/or alkaline phosphatase >2x upper limit of normal (ULN). Retesting is allowed once.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (18):
- United States (7):
  - Pacific Arthritis Care Center, Los Angeles, California
  - UCLA Rheumatology, Los Angeles, California
  - RASF Clinical Research Center, Boca Raton, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Metroplex Clinical Research Center, Dallas, Texas
  - UT Physicians Center for Autoimmunity, Houston, Texas
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
- Italy (2):
  - Azienda Ospedaliero, Florence
  - Ospedale San Raffaele S.r.l. - PPDS, Milan
- Spain (3):
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Nuestra Señora de Valme, Seville
- United Kingdom (2):
  - University Hospital Aintree, Liverpool
  - Royal Free Hospital, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Belgium, the United States, United Kingdom, Spain, and Italy. The first participant was screened on 14 Jan 2019. The last study visit occurred on 22 Jun 2020.
Pre-assignment Details: A total of 40 participants were screened, of whom 33 participants were randomized and treated.
Period: Overall Study
Arm/Group | GLPG1690 600 mg | Placebo
Started | 21 | 12
Completed | 21 | 11
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) consisted of all randomized participants who received at least 1 dose of investigational product.
Groups:
- GLPG1690 600 mg: Participants received GLPG1690 600 mg, orally once daily for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | GLPG1690 600 mg | Placebo | Total
Number analyzed (Participants) | 21 | 12 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (13.58) | 47.3 (17.99) | 49.3 (15.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 8 | 23
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 10 | 30
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 11 | 32
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Modified Rodnan Skin Score (mRSS) [Mean (Standard Deviation); unit: units on a scale] — The mRSS is a validated physical examination method for estimating skin thickness. The 17 body site mRSS was used, with each body site assessed on a scale of 0 (uninvolved) to 3 (severe thickening) with a total score range from 0 (best) to 51 (worst), with higher scores indicating greater severity of skin thickening.
  units on a scale | 27.0 (8.84) | 22.5 (6.24) | 25.3 (8.18)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in mRSS at Week 4
Description: The mRSS is a validated physical examination method for estimating skin thickness. The 17 body site mRSS was used, with each body site assessed on a scale of 0 (uninvolved) to 3 (severe thickening) with a total score range from 0 (best) to 51 (worst), with higher scores indicating greater severity of skin thickening.
Time Frame: Baseline, Week 4
Population: Participants in the FAS were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | GLPG1690 600 mg | Placebo
Number analyzed (Participants) | 21 | 12
units on a scale | -2.2 (0.85) | -1.6 (1.04)
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; Results were estimated using a mixed-effect model repeated measure using treatment and visit as fixed effects, baseline mRSS score and country as covariates, treatment-visit as interaction terms, and participant as a random effect. The variance-covariance matrix used in the model was compound symmetric; Test type: Superiority; p = 0.6757, Mixed Models Analysis; Least square (LS) mean difference = -0.5, 95% CI 2-sided [-3.1 to 2.0], Standard Error of Mean 1.29 — A negative difference indicates a greater improvement in the GLPG1690 treatment group

2. Primary Outcome: Change From Baseline in mRSS at Week 8
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: Participants in the FAS were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | GLPG1690 600 mg | Placebo
Number analyzed (Participants) | 21 | 12
units on a scale | -3.2 (0.85) | -2.5 (1.07)
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6079, Mixed Models Analysis; LS mean difference = -0.7, 95% CI 2-sided [-3.3 to 1.9], Standard Error of Mean 1.31 — A negative difference indicates a greater improvement in the GLPG1690 treatment group

3. Primary Outcome: Change From Baseline in mRSS at Week 16
Description: as for outcome 1
Time Frame: Baseline, Week 16
Population: Participants in the FAS were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | GLPG1690 600 mg | Placebo
Number analyzed (Participants) | 21 | 12
units on a scale | -6.8 (0.85) | -4.8 (1.12)
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1298, Mixed Models Analysis; LS mean difference = -2.1, 95% CI 2-sided [-4.8 to 0.6], Standard Error of Mean 1.35 — A negative difference indicates a greater improvement in the GLPG1690 treatment group

4. Primary Outcome: Change From Baseline in mRSS at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: Participants in the FAS were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | GLPG1690 600 mg | Placebo
Number analyzed (Participants) | 21 | 12
units on a scale | -8.9 (0.87) | -6.0 (1.11)
Statistical Analysis 1: Comparison: GLPG1690 600 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0411, Mixed Models Analysis; LS mean difference = -2.8, 95% CI 2-sided [-5.6 to -0.1], Standard Error of Mean 1.36 — A negative difference indicates a greater improvement in the GLPG1690 treatment group

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered study drug and which did not necessarily have a causal relationship with study drug. A treatment-emergent adverse event (TEAE) is any AE with an onset date on or after the start of stud drug intake and no later than 30 days after last dose of study drug, or any worsening of any AE on or after the start of stud drug intake. A serious AE was defined as an AE that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was medically significant.
Time Frame: Baseline up to end of the study (36 weeks)
Population: Safety analysis set consisted of all randomized participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | GLPG1690 600 mg | Placebo
Number analyzed (Participants) | 21 | 12
Participants
  TEAEs | 20 | 11
  Serious TEAEs | 2 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to end of the study (36 weeks)
Description: Participants in the safety analysis set were analyzed.
Arm/Group | GLPG1690 600 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/21 | 1/12
Other Adverse Events (participants affected / at risk) | 20/21 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GLPG1690 600 mg (N=21) | Placebo (N=12)
Sepsis (Infections and infestations) | 2 | 0
Device related infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GLPG1690 600 mg (N=21) | Placebo (N=12)
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Rhinitis (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Suspected COVID-19 (Infections and infestations) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Eructation (Gastrointestinal disorders) | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gingival recession (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 2
Dizziness (Nervous system disorders) | 3 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 0
Digital pitting scar (Skin and subcutaneous tissue disorders) | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Vascular injury (Injury, poisoning and procedural complications) | 1 | 0
Peripheral swelling (General disorders) | 3 | 0
Discomfort (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Palpitations (Cardiac disorders) | 2 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Weight increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Anger (Psychiatric disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Hot flush (Vascular disorders) | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
This was a proof-of-concept study not sized or powered to confirm any treatment effect.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review and approve any results of the study or abstracts for professional meetings prepared by the investigator(s). Published data must not compromise the objectives of the study. Data from individual study centers in multicenter studies must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT03798366/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT03798366/SAP_001.pdf